CLINICAL TRIAL: NCT04683861
Title: Spinal Cord Stimulation Therapy for Freezing of Gait in Patients With Advanced Parkinson's Disease and Parkinsonism-Plus Syndrome
Brief Title: Spinal Cord Stimulation Therapy for Freezing of Gait in Parkinson's Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: zhangyuqing (Other)
Responsible Party: Sponsor-Investigator, zhangyuqing, Clinical Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201203
Record Dates: First submitted 2020-12-03; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Freezing of Gait
Keywords: spinal cord stimulation; freezing of gait; Parkinson's disease; Parkinsonism-Plus syndrome
MeSH Terms: conditions — Parkinson Disease | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord stimulation therapy (Experimental): Spinal cord stimulation at the thoracic levels ranging from T10 to T12.
  Interventions: Procedure: Spinal cord stimulation

INTERVENTIONS:
Procedure: Spinal cord stimulation — Paddle-shaped Spinal cord stimulation electrode with 16 contacts (AdaptiveStim® 39, 565; Medtronic, USA) will be implanted into the epidural space at the thoracic levels ranging from T10 to T12.

SUMMARY:
Spinal cord stimulation may be a new therapeutic approach for freezing of gait. It's a multi-center, prospective, open label clinical study with a 12 months follow-up period, to investigate the therapeutic effect and safety of spinal cord stimulation for freezing of gait in patients with advanced Parkinson's disease and Parkinsonism-Plus syndrome.

DETAILED DESCRIPTION:
Benefits of dopaminergic therapy and deep brain stimulation are limited for freezing of gait in Parkinson's syndrome. Spinal cord stimulation is a well-established therapy for the treatment of chronic neuropathic pain. Recently, some pilot studies demonstrated the safety and significant therapeutic effect of Spinal cord stimulation in freezing of gait patients suffering from various movement disorders, such as Parkinson's disease, primary progressive freezing of gait, and multiple system atrophy with predominant Parkinsonism. Spinal cord stimulation may be a new therapeutic approach for freezing of gait. However, evidence from larger numbers of subjects is still lacking, especially little is known about its efficacy for gait and posture dysfunction in Parkinsonism-Plus syndrome patients. The objective of this study is to investigate the therapeutic effect and safety of spinal cord stimulation for freezing of gait in patients with advanced Parkinson's disease and Parkinsonism-Plus syndrome.

It's a multi-center, prospective, open label clinical study with a 12 months follow-up period. The intended study population is individuals suffering from advanced Parkinson's disease, multiple system atrophy with predominant parkinsonism or progressive supranuclear palsy. Each participant will complete an enrollment/screening/baseline visit, a spinal cord stimulation implant and activation visit, and a minimum of two follow-up visits, including visit at 3 months and the final study visit at 12months. The participants will proceed to implantation after satisfying implant inclusion and exclusion criteria. Paddle-shaped Spinal cord stimulation electrode with 16 contacts (AdaptiveStim® 39, 565; Medtronic, Minneapolis, USA) will be implanted into the epidural space at the thoracic levels ranging from T10 to T12. Electrode position will be verified by X-ray. The stimulators will be turned on within 1 month after electrode implantation surgery. The stimulation parameters could vary freely, but medications will be kept constant during the study period. At the end of month 12, participants will enter the long-term follow-up in which medications and stimulation parameters could vary freely.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 40 and 76 years
2. patients with advanced Parkinson's disease, or multiple system atrophy with predominant parkinsonism or progressive supranuclear palsy (PSP)
3. with significant freezing of gait ( Movement Disorder Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale III item 11≥2), and the gait dysfunction treatable by medication but not adequately controlled with medications.
4. Understand potential risk/benefit, consent to the study, study procedures, and agree to complete the study follow-up visits and comply with the study protocol requirements.

Exclusion Criteria:

1. cognitive impairment ( MMSE≤24), depression (HAMD>24),acute psychosis, active alcohol or drug abuse, terminal illness, and any major medical or psychological histories, diagnoses, conditions, or comorbidities that would interfere with participation in the study per the investigatior's medical judgment
2. surgical or medical contraindications to spinal cord stimulation surgery(e.g. uncontrolled hypertension, advanced coronary artery disease).

Ages: 40 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
change in severity of freezing of gait | twelve months after surgery
  demonstrate statistically significant improvement in score of "New Freezing of Gait Questionnaire (NFOGQ)" from baseline to 12 months
change in the score of "Gait and Fall Questionnaire (GFQ)" | twelve months after surgery.
  demonstrate statistically significant improvement in score of GFQ from baseline to 12 months

SECONDARY OUTCOMES:
change in PD-related quality of life(PDQ-39) | twelve months after surgery.
  demonstrate statistically significant improvement in PD-related quality of life(PDQ-39) from baseline to 12 months
change in motor examination( Movement Disorders Society's revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III) | twelve months after surgery.
  demonstrate the change in motor score (MDS-UPDRS III) from baseline( Off medication) to 12 months (On stimulation/Off medication)
Clinical Global Impression-Global Improvement (CGI-GI) | twelve months after surgery.
  to evaluate effectiveness on the basis of the physician's assessment, as well as on the basis of the patients'self-reported satisfaction. It is rated on a 7-point scale, range from 1(very much improved) through to 7 (very much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Yuqung Zhang, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Capital Medical University of Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No